CLINICAL TRIAL: NCT02908659
Title: Relevance and Possible Nuisances of Respiratory Rate Alarm Generated by Multi-parametric Monitors in Non Ventilated ICU Patients.A Prospective, Monocentric, Observational Study
Brief Title: Relevance and Nuisances of Respiratory Rate Alarm Generated by Multi-parametric Monitors in Non Ventilated ICU Patients
Acronym: FR-REA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD 087-16
Record Dates: First submitted 2016-09-07; First posted 2016-09-21 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Non Ventilated ICU Patients
Keywords: intensive care unit; patient's monitoring; respiratory rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In ICU setting, a large number of medical devices are attached to patients, generating numerous alarm signals. Several studies have demonstrated that most of these alarms are not clinically relevant and tend to lower the attentiveness of healthcare professional and, in turn, lower patient safety.The aim of the study is to assess the relevance of respiratory rate alarm on a monitoring device in non-ventilated ICU patients.

The investigator primary hypothesis is that this alarm is potentially useless. If this hypothesis is confirmed, a second interventional trial will be conducted on the impact of this alarm removal.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patient hospitalized in ICU
* Need for monitoring

Exclusion Criteria:

* Invasive mechanical ventilation
* Non-invasive mechanical ventilation
* Patient not monitored
* Patient already included in this study
* Patient hospitalized without consent and/or deprived of liberty by court's decision
* Patient under guardianship or curators
* Lack of social insurance
* Patient's or next of kin's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU unit at La Roche sur yon Hospital
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Number of useful alarms within 2000 patient-monitored hours | through study completion, within 6 months
  Number of intervention of healthcare team following a relevant respiratory rate alarm generated by a monitoring device and without any other associated alarm.

SECONDARY OUTCOMES:
Ratio of artifact alarms among all alarms generated by the monitoring device | through study completion within 6 months
  Artifact alarm : monitoring is functional but the measure is false
Ratio of technical alarms among all alarms generated by the monitoring device | through study completion within 6 months
  Technical alarm : Alarm leading to a reactivation of the monitoring system.
Ratio of significant alarms among all alarms generated by the monitoring device | through study completion within 6 months
  Significant alarm: True alarm triggered by a correct measure
Number of care activity interrupted by a respiratory rate alarm generated by the monitoring device | through study completion within 6 months
Setting of alarms on the monitoring device | through study completion within 6 months
ICU length of stay | Until discharge from ICU, an expected average of 7 days
all-cause ICU mortality | Until discharge from ICU, an expected average of 7 days ]
Ratio of respiratory rate alarms generated by the monitoring device among all ICU alarms | through study completion within 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHD Vendee, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No